CLINICAL TRIAL: NCT01344213
Title: Comparison of Analgesic Efficacy Among Pregabalin, Celecoxib, Pregabalin With Celecoxib and Placebo After Total Knee Arthroplasty Under Intrathecal Morphine
Brief Title: Pregabalin, Celecoxib, Total Knee Arthroplasty and Intrathecal Morphine
Acronym: PCTKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Bhumibol Adulyadej Hospital (Other); King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Assoc.Professor Supranee Niruthisard, Department of Anesthesiology, Faculty of Medicine, Chulalongkorn Unv.
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: anesTKA08
Record Dates: First submitted 2011-04-26; First posted 2011-04-29 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-04

CONDITIONS: Postoperative Pain Management; Total Knee Arthroplasty
Keywords: Pregabalin; Celecoxib; Intrathecal morphine; Total knee arthroplasty
MeSH Terms: interventions — Pregabalin; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Pregabalin (Active Comparator): Oral single-dose of pregabalin (150 mg) and 1 capsule of placebo (P) 1-2 hours before starting spinal anesthesia with intrathecal morphine 0.2 mg.
  Interventions: Drug: Pregabalin
- Celecoxib (Active Comparator): Oral single-dose of celecoxib (400 mg) and 1 capsule of placebo (C) 1-2 hours before starting spinal anesthesia with intrathecal morphine 0.2 mg.
  Interventions: Drug: Celecoxib
- Pregabalin with celecoxib (Active Comparator): Oral single-dose of pregabalin (150 mg) and celecoxib (400 mg) (PC) 1-2 hours before starting spinal anesthesia with intrathecal morphine 0.2 mg.
  Interventions: Drug: Pregabalin with celecoxib
- Placebo (Placebo Comparator): Oral single-dose of placebo 2 capsules 1-2 hours before starting spinal anesthesia with intrathecal morphine 0.2 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Oral single-dose of pregabalin (150 mg) and placebo (P) 1-2 hours before starting spinal anesthesia with intrathecal morphine 0.2 mg.
  Other Names: Pregabalin: Lyrica
  Arms: Pregabalin
Drug: Celecoxib — Oral single-dose of celecoxib (400 mg) and placebo(C)1-2 hours before starting spinal anesthesia with intrathecal morphine 0.2 mg.
  Other Names: Celecoxib: Celebrex
  Arms: Celecoxib
Drug: Pregabalin with celecoxib — Oral single-dose of pregabalin (150 mg) and celecoxib (400 mg) (PC) 1-2 hours before starting spinal anesthesia with intrathecal morphine 0.2 mg.
  Other Names: Pregabalin: Lyrica; Celecoxib: Celebrex
  Arms: Pregabalin with celecoxib
Drug: Placebo — Oral single dose of placebo 2 capsules 1-2 hours before starting spinal anesthesia with intrathecal morphine 0.2 mg
  Other Names: Placebo: sugar capsule
  Arms: Placebo

SUMMARY:
To evaluate whether pregabalin and/or celecoxib could improve analgesic efficacy of intrathecal morphine for patients after total knee arthroplasty.

DETAILED DESCRIPTION:
A single-dose spinal anesthesia combining with morphine for total knee arthroplasty (TKA) is a simple, economical anesthetic technique commonly used in our hospital. Still some patients could not get effective postoperative pain control. Pregabalin, an anticonvulsant, has been shown to reduce acute pain after molar extraction, laparoscopic cholecystectomy, and reduce postoperative morphine requirement after total hip arthroplasty, and celecoxib, a selective cyclo-oxygenase (COX) - 2 inhibitor, with perioperative prescription is successfully reduces pain score and opioid consumption after TKA under spinal anesthesia alone. However, no clinical study has yet investigated whether preoperative single-dose of pregabalin, celecoxib or in combination compared to placebo can improve analgesic efficacy of intrathecal morphine after TKA. The primary objective of this study was to evaluate whether these medications could reduce pain scores at rest / when movement and morphine requirement after TKA under spinal anesthesia with intrathecal morphine. Secondary outcome assessed include adverse effects, anxiety score and patients' satisfaction score.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 50-75 years of age
* Patients with an American Society of Anesthesiologists physical status of I to III
* Patients scheduled for primary TKA with a diagnosis of osteoarthritis under spinal anesthesia

Exclusion Criteria:.

* Patients had a known allergy to any of the medications being used
* a history of drug or alcohol abuse
* a history of taking chronic pain medications (ie, show-release preparations of opioids, given that morphine consumption was the primary outcome)
* a history of taking pregabalin or gabapentin / non-steroidal anti-inflammatory drugs / COX-2 inhibitors
* a psychiatric disorder
* a history of impaired renal function (Cr > 1.5 mg/dl), peptic ulcer, asthma, thrombotic cerebrocardiovascular diseases, uncontrolled hypertension
* a history of contraindication for spinal anesthesia
* a history of bleeding tendency
* pregnancy
* unable or unwilling to use patient - controlled analgesic (PCA)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-07; Primary Completion 2009-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
24-hour cumulative morphine consumption | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  * The time to first morphine requirement will be recorded
  * The cumulative morphine consumption will be recorded at the end of surgery and 2-h, 6-h, 10-h, 24-h, and 48-h postoperatively
  * Visual analog scale (VAS) pain scores at rest will be assessed at the night before surgical date, before starting anesthesia, at the end of surgery, and 2-h, 6-h, 10-h, 24-h and 48-h postoperatively
  * Visual analog scale (VAS) pain scores when on movement will be assessed at the end of surgery, and 2-h, 6-h, 10-h, 24-h and 48-h postoperatively

SECONDARY OUTCOMES:
Anxiety scores (VAS), patients' satisfaction | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  * Anxiety scores will be assessed at the night before surgical date, before starting anesthesia, at the end of surgery, and 2-h, 6-h, 10-h, 24-h and 48-h postoperatively;
  * 24-h and 48-h patients' satisfaction (0-10,0=dissatisfied and 10= very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Supranee Niruthisard, BSc, MD, Principal Investigator — King Chulalongkorn Memorial Hospital
Locations (1):
- Supranee Niruthisard, Bangkok, Thailand